CLINICAL TRIAL: NCT05234840
Title: "Platelet-Rich Plasma" Transforaminal Epidural Injection an Emerging Strategy in Lumbar Disc Herniation
Brief Title: "Platelet-Rich Plasma" Epidural Injection an Emerging Strategy in Lumbar Disc Herniation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Savang Vadhana Memorial Hospital, Thailand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 015/2563
Record Dates: First submitted 2022-01-10; First posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: PRP
Keywords: PRP, HNP, lumbar HNP
MeSH Terms: interventions — Triamcinolone

STUDY DESIGN:
Intervention Model Description: Thirty patients were treated by transforaminal epidural injections. Fifteen patients were in triamcinolone and PRP groups each. PRP was obtained from 24 ml venous blood through standardized double-spin protocol. Participants were fifteen patients each in triamcinolone and PRP groups. The same postoperative protocols and medications were applied. The visual analogue scale of leg (LegVAS), collected at baseline, 2, 6, 12, and 24 weeks, was the primary outcome.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: all patient were masked. Surgeon was blinded by leukostrip around injection syringe. Assessor was blinded from operative information.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Triamcinolone group (Active Comparator): Patients were placed in the prone position. Transforaminal triamcinolone injections were performed under a C-arm fluoroscopy.
  Interventions: Drug: Triamcinolone
- Platelet-rich plasma (Experimental): Patients were placed in the prone position. Transforaminal PRPinjections were performed under a C-arm fluoroscopy.
  Interventions: Drug: platelet rich plasma

INTERVENTIONS:
Drug: platelet rich plasma — 1. 26 ml of blood was obtained from each patient (6ml each in 4 CPDA and 2ml in EDTA for CBC) 2. First-spin of 900g for 5 minutes (Kokusan, H-19alpha, 25°C) 3. Three layers formed: transfer top layer (platelet poor plasma) and middle layer (platelets and WBC) to another sterile tube (about 3.3 ml), discard bottom layer (RBC) 4. Second-spin of 1000g for 10 minutes 5. The upper one third was discarded (platelet poor plasma) by pipet, the remaining was mixed by turning 10 times 6. Total 4 ml of PRP
  Other Names: PRP
  Arms: Platelet-rich plasma
Drug: Triamcinolone — 40 mg triamcinolone with 1% lidocaine, total of 2 ml
  Other Names: kenacort
  Arms: Triamcinolone group

SUMMARY:
To evaluate the efficacy of platelet-rich plasma (PRP; double-spin) in treatment of single-level lumbar herniated nucleus pulposus (HNP) in comparison to triamcinolone. RCT was conducted with 30 patients included.

DETAILED DESCRIPTION:
The study was a randomized controlled trial, triple-blind, single-center/surgeon/assessor. The study was conducted between April 2019 to May 2021. We evaluated 30 patients (both genders) aged 20-55 years, having failed conservative treatment of unilateral HNP undergone for at least 6 weeks, with visual analogue scale (VAS) of greater than 30, and confirmed a single-level HNP, corelated to clinical, by MRI. The exclusion criteria included previous spine surgery or epidural injection, progressive neurological deficit, cauda equina, coagulopathy-related conditions, associated cervical myelopathy, systemic bone and joint diseases. All patients had to have been exempted from NSAIDs for at least one week. Patients were treated by transforaminal epidural injections. Fifteen patients were in triamcinolone and PRP groups each. PRP was obtained from 24 ml venous blood through standardized double-spin protocol. Participants were fifteen patients each in triamcinolone and PRP groups. The same postoperative protocols and medications were applied. The visual analogue scale of leg (LegVAS), collected at baseline, 2, 6, 12, and 24 weeks, was the primary outcome. The BackVAS, Oswestry Disability Index (ODI), adverse event, and treatment failure were the secondary endpoints. All subjects were analyzed according to the intention-to-treat principle. All statistical analyses were performed with STATA 17.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-55 years
* Having failed conservative treatment for at least 6 weeks
* Visual analogue scale (VAS) of greater than 30
* Confirmed a single-level HNP, corelated to clinical, by MRI.

Exclusion Criteria:

* Previous spine surgery or epidural injection
* Progressive neurological deficit
* Cauda equina
* Coagulopathy-related conditions
* Associated cervical myelopathy
* Systemic bone and joint diseases

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
VAS of leg pain | at 24 weeks
  0-100 (visual analog score, 0 is the minimum and 100 is the maximum)

SECONDARY OUTCOMES:
VAS of back | at 24 weeks
  0-100 (visual analog score, 0 is the minimum and 100 is the maximum)
ODI | at 24 weeks
  Oswestry Disability Index 0-100% (0 is the minimum and 100 is the maximum)
adverse event | up to 24 weeks
  minor and major complications from injection
Rate of treatment failure [participant who require reinjection or operation] | up to 24 weeks
  During follow-up period, participant require either re-injection or operation [yes/no]

CONTACTS AND LOCATIONS:
Locations (1):
- Chuenrutai, Chon Buri, Thailand

IPD SHARING:
Plan to Share IPD: Undecided
Data was save in form of Microsoft excel spreadsheet and STATA file.

REFERENCES:
- [Background] Dhurat R, Sukesh M. Principles and Methods of Preparation of Platelet-Rich Plasma: A Review and Author's Perspective. J Cutan Aesthet Surg. 2014 Oct-Dec;7(4):189-97. doi: 10.4103/0974-2077.150734. PMID 25722595
- [Background] Becker C, Heidersdorf S, Drewlo S, de Rodriguez SZ, Kramer J, Willburger RE. Efficacy of epidural perineural injections with autologous conditioned serum for lumbar radicular compression: an investigator-initiated, prospective, double-blind, reference-controlled study. Spine (Phila Pa 1976). 2007 Aug 1;32(17):1803-8. doi: 10.1097/BRS.0b013e3181076514. PMID 17762286
- [Background] Centeno C, Markle J, Dodson E, Stemper I, Hyzy M, Williams C, Freeman M. The use of lumbar epidural injection of platelet lysate for treatment of radicular pain. J Exp Orthop. 2017 Nov 25;4(1):38. doi: 10.1186/s40634-017-0113-5. PMID 29177632
- [Background] Cameron JA TK. Autologous Platelet Rich Plasma for Neck and Lower Back Pain Secondary to Spinal Disc Herniation: Midterm Results. Spine Res 2017;32.
- [Background] H S RK, Goni VG, Y K B. Autologous Conditioned Serum as a Novel Alternative Option in the Treatment of Unilateral Lumbar Radiculopathy: A Prospective Study. Asian Spine J. 2015 Dec;9(6):916-22. doi: 10.4184/asj.2015.9.6.916. Epub 2015 Dec 8. PMID 26713125
- [Derived] Wongjarupong A, Pairuchvej S, Laohapornsvan P, Kotheeranurak V, Jitpakdee K, Yeekian C, Chanplakorn P. "Platelet-Rich Plasma" epidural injection an emerging strategy in lumbar disc herniation: a Randomized Controlled Trial. BMC Musculoskelet Disord. 2023 Apr 28;24(1):335. doi: 10.1186/s12891-023-06429-3. PMID 37118707